CLINICAL TRIAL: NCT06691815
Title: Early Diagnosis of Hypogonadotrophic Hypogonadism by a Gonadotrophic-gonadal Stimulation Test with GnRH Agonist (Triptorelin)
Brief Title: Triptorelin for Early Diagnosis of Hypogonadotrophic Hypogonadism
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Analía Freire, Principal investigator, Hospital de Niños R. Gutierrez de Buenos Aires
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hospital de Niños R. Gutierrez; CEI 22.23 (Other: Ethics Committee of the Hospital de Niños Dr. Ricardo Gutiérrez)
Record Dates: First submitted 2024-10-23; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Pubertal Delay; Hypogonadism, Hypogonadotropic; Constitutional Delay in Growth and Puberty (CDGP)
Keywords: Hypogonadism, hypogonadotropic; Constitutional Delay in Growth and Puberty; Pubertal Delay; GnRH agonist test; Gondotropins; gonadal steroids
MeSH Terms: conditions — Puberty, Delayed; Hypogonadism

STUDY DESIGN:
Intervention Model Description: The order in which the tests will be performed will be randomized at the time the patients are included in the study.
  1. Triptorelin test. A baseline blood sample will be taken to determine LH, FSH, Estradiol/Testosterone, AMH, and Inhibin B. Then, Triptorelin Acetate 100 ug/m² of body surface area will be administered subcutaneously, maximum dose 0.1 mg (Decapeptyl Daily prefilled syringe of 0.1 mg for subcutaneous administration. Three hours later, a new sample will be taken to determine LH and FSH. The patient may return home and lead a normal life. An appointment will be made the following day to perform the last sample of this test 24 hours after the subcutaneous administration of Triptorelin Acetate, with the determination of LH, FSH, Estradiol/Testosterone, and Inhibin B.
  2. GnRH Infusion: This consists of determining LH and FSH in baseline blood samples, 15, 30, 45, 60 and 120 minutes after slow infusion of GnRH. GnRH 0.83 μg/min during the 120 minutes that the study lasts (Lu
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Unique arm (Experimental): All patients will be randomized only to the order of the test to be performed. All patients included will be performed two tes
  1. Triptorelin test. A baseline blood sample will be taken to determine LH, FSH, Estradiol/Testosterone. Then, Triptorelin Acetate 100 ug/m² of body surface area will be administered subcutaneously, maximum dose 0.1 mg (Decapeptyl Daily prefilled syringe of 0.1 mg) Three hours later, a new sample will be taken to determine LH and FSH. The patient may return home and lead a normal life. An appointment will be made the following day to perform the last sample of this test 24 hours after the subcutaneous administration of Triptorelin to the meassurement of LH, FSH, Estradiol/Testosterone, and Inhibin B.
  2. GnRH Infusion: LH and FSH in baseline blood samples, 15, 30, 45, 60 and 120 minutes after slow infusion of GnRH. GnRH 0.83 μg/min during the 120 minutes that the study lasts (Luteoliberin 100 μg)
  Interventions: Diagnostic Test: Triptorelin (GnRH agonists)

INTERVENTIONS:
Diagnostic Test: Triptorelin (GnRH agonists) — 1. Triptorelin test. A baseline blood sample will be taken to determine LH, FSH, Estradiol/Testosterone, AMH, and Inhibin B. Then, Triptorelin Acetate 100 ug/m² of body surface area will be administered subcutaneously, maximum dose 0.1 mg (Decapeptyl Daily prefilled syringe of 0.1 mg for subcutaneous administration. Three hours later, a new sample will be taken to determine LH and FSH. The patient may return home and lead a normal life. An appointment will be made the following day to perform the last sample of this test 24 hours after the subcutaneous administration of Triptorelin Acetate, with the determination of LH, FSH, Estradiol/Testosterone, and Inhibin B.
  2. GnRH Infusion: This consists of determining LH and FSH in baseline blood samples, 15, 30, 45, 60 and 120 minutes after slow infusion of GnRH. GnRH 0.83 μg/min during the 120 minutes that the study lasts (Luteoliberin 100 μg)
  Other Names: Triptorelin 0.1 mg subcutaneos test

SUMMARY:
The goal of this clinical trial is to learn if Triptorelin test works to early diagnose hypogonadotrophic hypogonadism in adolescents. The main questions it aims to answer are:

• Does gonadotropin and gonadal steroids responses to Triptorelin test be useful to diagnose early hypogonadotrophic hypogonadism? Researchers will compare gonadotrophins and gonadal steroids in response to Triptorelin subucutaneos test with clasiccal GnRH infusion to diagnose hypogonadotrophic hypogonadism.

Participants will performed two test:

* Triptorelin test (subcutanous)
* LHRH infusion test

ELIGIBILITY:
Inclusion Criteria:

* Female patients presenting with Tanner breast stage 1 or 2 at age ≥ 13 years or male patients with testicular volume < 5 cc at age ≥ 13.5 years, or who have had pubertal changes but have arrested pubertal development for a period of one year. Female patients presenting with primary amenorrhea (absence of menarche at age 15) > 4 years after the onset of puberty or secondary amenorrhea > 6 months with no other apparent cause (having ruled out other hormonal disorders such as premature ovarian failure, hypothyroidism, hyperprolactinemia, non-classical congenital adrenal hyperplasia, and polycystic ovary syndrome) may also be included. Patients with or without olfactory disorders, and with or without a previous diagnosis of other pituitary deficiencies will be included. In the case of a history of CNS tumor pathology, inclusion in this study will be considered only if the patient is in remission from the oncological disease and if they have received CNS radiotherapy, at least one year has passed since the beginning of the treatment.

If patients have started HRT, they may be included as long as they stop taking it for two half-lives of the compound used, therefore a 2-month free period is necessary for oral tablets or patches and 3 months for monthly testosterone injections or 7 months for testosterone undecanoate injections.

Exclusion Criteria:

* Patients will be excluded if, due to previous history or relevant clinical history or initial laboratory study, another cause is determined to explain their pubertal disorder: primary hypogonadism (hypergonadotrophic or premature ovarian failure), low weight with BMI < 18, untreated hypothyroidism, hyperprolactinemia, hyperandrogenism, Cushing's syndrome, current prolonged corticosteroid treatment, active systemic disease, CRF or competitive training > 10 hours/week, diabetes mellitus without adequate control or celiac disease without compliance with a gluten-free diet.

Patients who do not provide an updated medical history, who do not provide consent, or whose parents or guardians do not provide assent will be excluded. Patients who are receiving hormone replacement therapy and refuse to stop during the 2-month period for oral tablets or patches and 3 months for monthly testosterone injections or 7 months for quarterly depot injections of testosterone undecanoate will be excluded.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
LH-3 hs, FSH-3 hs, Estradiol-24 hs, Testosteron-24 hs | -To finish spontanous puberty or to get the definitive diagnosis of hypogonadotrophic hypogonadism
  LH, FSH, Estradiol or Testosterone meassurement in samples 3 hs o 24 hs after triptorelin subcutaneous administration

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Niños Dr. Ricardo Gutiérrez, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided